CLINICAL TRIAL: NCT03847155
Title: Prevention of Nicotine Abstinence in Critically Ill Patients After Major Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Ostrava (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: KARIM-09-NICOTINE; 2014-003720-43 (EudraCT Number)
Record Dates: First submitted 2019-02-18; First posted 2019-02-20 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Nicotine Dependence
Keywords: nicotine patch; placebo; critically ill patients; delirium; prevention
MeSH Terms: conditions — Tobacco Use Disorder; Delirium | interventions — Tobacco Use Cessation Devices

STUDY DESIGN:
Intervention Model Description: The patients will be randomized into two study groups, with the active substance and placebo.
Who Masked: Participant, Care Provider, Investigator
Masking Description: The participant, care provider and investigator will be masked as far as the treatment provided is concerned.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nicotine (Experimental): The patients randomized into this study arm will receive a medical intervention - nicotine patch for the period of a maximum of 7 days.
  Interventions: Drug: Nicotine patch
- Placebo (Placebo Comparator): The patients randomized into this study arm will receive a placebo patch for the period of a maximum of 7 days.
  Interventions: Other: Placebo patch

INTERVENTIONS:
Drug: Nicotine patch — The patients will receive a nicotine patch for the period of a maximum of 7 days.
  Arms: Nicotine
Other: Placebo patch — The patients will receive a placebo patch for the period of a maximum of 7 days.
  Arms: Placebo

SUMMARY:
The primary objective of this study is to determine whether the application of transdermal nicotine patches in critically ill patients after major surgery with nicotine abstinence condition is associated with a lower incidence of delirium.

DETAILED DESCRIPTION:
Patients in a group with medical intervention receive nicotine patch within 24 hours after surgery. The nicotine patch is replaced every day. Delirium is evaluated every day by the Confusion Assessment Method (CAM) - ICU test. The maximum length of intervention is 7 days.

Patients in a group with placebo receive a placebo patch within 24 hours after surgery. This patch is replaced every day. Delirium is evaluated in the same way - CAM - ICU test. The maximum length of the placebo intervention is 7 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing a surgical procedure - urological, surgical, trauma surgery, orthopedic surgery, dental surgery)
* Age 18 years and above
* Patient with an assumption of nicotine abstinence (smoking a minimum 10 cigarettes/day).
* Ex-smokers (if they stopped smoking less than 30 days prior to surgery)
* An assumption of hospitalization at the intensive care unit (ICU) after surgery
* Signed Informed consent

Exclusion Criteria:

* Age ˂ 18 years
* Non-signing of the informed consent
* Patients after neurosurgical surgery, patients with traumatic brain injury, patients after a new stroke
* Patients with psychiatric diseases
* Nicotine, Curapor or Hydrocoll allergy
* Patient with a heart attack, unstable angina pectoris or patients with a serious heart arrhythmia
* Pregnant and breastfeeding patients
* Patients with nicotine treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2015-09-23 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-02-08 (Actual)

PRIMARY OUTCOMES:
Incidence of delirium episodes | maximum of 7 days
  The number of delirium episodes, defined according to the CAM-ICU test, in the course of the seven days with the patch attached will be measured in both groups of study subjects.

SECONDARY OUTCOMES:
Change in the number of days with delirium | maximum of 7 days
  Change in the number of days with delirium, defined according to the CAM-ICU test, by 20%, in the course of the seven days with the patch attached among the study subjects with the nicotine patch.
Ventilator-hours | maximum of 7 days
  The number of ventilator-hours will be observed in both groups of study subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Neiser, MD, Principal Investigator — University Hospital Ostrava
Locations (1):
- University Hospital Ostrava, Ostrava, Moravian-Silesian Region, Czechia

IPD SHARING:
Plan to Share IPD: No
The investigators do not plan to make individual participant data available to other researchers.

REFERENCES:
- [Background] Granberg Axell AI, Malmros CW, Bergbom IL, Lundberg DB. Intensive care unit syndrome/delirium is associated with anemia, drug therapy and duration of ventilation treatment. Acta Anaesthesiol Scand. 2002 Jul;46(6):726-31. doi: 10.1034/j.1399-6576.2002.460616.x. PMID 12059899
- [Background] Bledowski J, Trutia A. A review of pharmacologic management and prevention strategies for delirium in the intensive care unit. Psychosomatics. 2012 May-Jun;53(3):203-11. doi: 10.1016/j.psym.2011.12.005. Epub 2012 Apr 4. PMID 22480622
- [Background] Cartin-Ceba R, Warner DO, Hays JT, Afessa B. Nicotine replacement therapy in critically ill patients: a prospective observational cohort study. Crit Care Med. 2011 Jul;39(7):1635-40. doi: 10.1097/CCM.0b013e31821867b8. PMID 21494111
- [Background] Jablonski J, Gray J, Miano T, Redline G, Teufel H, Collins T, Pascual-Lopez J, Sylvia M, Martin ND. Pain, Agitation, and Delirium Guidelines: Interprofessional Perspectives to Translate the Evidence. Dimens Crit Care Nurs. 2017 May/Jun;36(3):164-173. doi: 10.1097/DCC.0000000000000239. PMID 28375992
- [Background] Van Rompaey B, Schuurmans MJ, Shortridge-Baggett LM, Truijen S, Elseviers M, Bossaert L. A comparison of the CAM-ICU and the NEECHAM Confusion Scale in intensive care delirium assessment: an observational study in non-intubated patients. Crit Care. 2008;12(1):R16. doi: 10.1186/cc6790. Epub 2008 Feb 18. PMID 18282269